CLINICAL TRIAL: NCT02824159
Title: Real Life Assessment of the Association and Its Determinants Between Side Effects and Plasmatic Concentrations of Two Protein Kinase Inhibitors: Ibrutinib (IMBRUVICA®) and Idelalisib (ZYDELIG®) in Hematological Malignancies Treatment.
Brief Title: Association Between Side Effects Occurrence and Concentrations of Ibrutinib and Idelalisib
Acronym: PK-E3I
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 15 7754 07; 2015-005572-17 (EudraCT Number)
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Hematological Malignancies
Keywords: ibrutinib; idelalisib; side effect; pharmacokinetic; plasma balance mean concentration
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Blood Specimen Collection; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples to be collected are :
  * Blood samples for dosage of drug in plasma (No DNA)
  * Blood samples (genetic profile of drug elimination and presence of treatment resistance mutation) and saliva samples (genetic profile drug elimination )
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with haematologic malignancies: Interventions to be administrated are :
  * Clinical examinations
  * Biological statement
  * Blood samples for pharmacokinetics exploration
  * Imagery with positron emission tomography scan or resonance magnetic imagery
  * Saliva samples for genetics analyses
  * Blood samples for treatment mutation resistance search
  * Quality of life scale questionary
  * Detection of adverse events
  Interventions: Other: Blood samples for pharmacokinetics exploration; Other: Imagery; Other: Quality of life scale; Other: Detection of adverse events; Genetic: Saliva samples; Genetic: Blood sample; Other: Biological statement; Other: Clinical examination

INTERVENTIONS:
Other: Blood samples for pharmacokinetics exploration — 6 blood sample at regular intervals
Other: Imagery — Efficacity will be assessed with 3 sessions of resonance magnetic imaging or positron emission tomography scan
Other: Quality of life scale — Quality of life will be evaluated with questionaries 5 times during the study
Other: Detection of adverse events — The detection will be assessed using the AMA (assistance des malades ambulatoires) system
Genetic: Saliva samples — Saliva samples will be collected to explore genetic characteristics of germinal DNA (genes involved in drug pharmacokinetic)
Genetic: Blood sample — A unique blood sample will be performed in order to determine characteristics of tumoral DNA (resistance to treatment mutation)
Other: Biological statement — The following parameters will be assessed :
  * Complete blood count
  * Hemoglobin
  * Hepatic enzymes
  * Creatinine clearance
  * Lactate dehydrogenase rate
  * Total bilirubin rate
  * Cluster of differentiation 4 T lymphocytes rate
  * Total gamma-globulins rate
Other: Clinical examination — The clinical examination are composed by :
  * Weigh, Height and body mass index measurement
  * Clinical state of patient during examination
  * Stage of the disease (OMS grade, binet classification, Ahn Arbor classification)
  * Presence of B symptomatology
  * Prognostic factors (Genetic, Mantle Cell Lymphoma International Prognostic Index, Follicular Lymphoma International Prognostic Index, presence of lymph nodes, other target organs ...)

SUMMARY:
Recently, European Medicines Agency approved ibrutinib and idelalisib to treat Chronic Lymphocytic Leukemia (CLL) and two lymphomas: Follicular Lymphoma (FL) for ibrutinib and Mantle cell lymphoma (MCL) for idelalisib.

Clinical trials for ibrutinib and idelalisib were performed with a small number of patients (300-350) and showed several side effects profiles. Since, pharmacokinetic properties of these 2 drugs highlight a interindividual variability of pharmacokinetic. The aim of this study is to determine the association between clinically significant side effects occurrence during the first year of treatment and plasma mean concentration of the steady state of ibrutinib or idelalisib at 1 month.

DETAILED DESCRIPTION:
Recently, European medicines agency approved ibrutinib and idelalisib in the treatment of Chronic Lymphocytic Leukemia (CLL) and two lymphomas: Follicular Lymphoma (FL) for ibrutinib and Mantle cell lymphoma (MCL) for idelalisib. Nevertheless, clinical trials for these two drugs were performed for only 300-350 patients and showed several side effects profiles, the most frequent were diarrhea, infection, cutaneous rash… For some patients, treatment had to be reduced or stopped temporary or definitely.

Pharmacokinetic properties of these two drugs highlight an interindividual pharmacokinetic considerable variability. The aim of this clinical research study is to determine the association between clinically significant side effects occurrence during the first year of treatment (serious adverse reaction and/or grade CTCAE ≥ 3 and/or leading a dosage concession) and plasma mean concentration of the steady state of ibrutinib or idelalisib performed at 1 month.

To determine plasma mean concentration of the steady state of ibrutinib or idelalisib, blood tests will be performed every scheduled monitoring at visit 1 month during a pharmacokinetic exploration and during scheduled medical consultation (2, 3, 6 and 12 months) and every unscheduled visit in case of side effect occurrence.

Every scheduled monitoring visit, blood tests will be performed to determine plasma concentration in drug. Complementary blood or salivary samples will be collected before the treatment, 24 months later and in case of relapse to determine genetic characteristics. In parallel, a logbook will be completed by the patient to collect side effects. Finally, an oncology certified nurse call patients every 2 weeks. In case of side effect occurrence a visit will be organized in the next 3 days and a blood test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Chronic Lymphocytic Leukaemia (CLL), or Follicular Lymphoma (FL) or Mantle cell lymphoma (MCL) and a first prescription of idelalisib or ibrutinib
* Patients must give written informed consent
* Patients with Health Insurance System

Exclusion Criteria:

* Patient who several blood tests can't be performed (poor venous access)
* Patients under legal guardian
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with haematologic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-04; Primary Completion 2020-11 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinically significant side effect occurence with plasma balance mean concentration in ibrutinib | 1 months after treatment initiation
  Plasma balance mean will be calculated with 6 blood samples collected at regular intervals during the visit
Evaluation of clinically significant side effect occurence with plasma balance mean concentration in idelalisib | 1 months after treatment initiation
  Plasma balance mean will be calculated with 6 blood samples collected at regular intervals during the visit

SECONDARY OUTCOMES:
Clinically significant side effect occurrence (Serious adverse reaction and/or grade CTCAE ≥ 3 and/or leading a dosage concession) as assessed by AMA (Assistance des Malades Ambulatoires) system | through the end of study (24 months)
Plasma balance mean concentration in ibrutinib with collection of blood samples | 1 month after inclusion
  Plasma balance mean will be calculated with 6 blood samples collected at regular intervals during the visit
Plasma balance mean concentration in idelalisib with collection of blood samples | 1 month after inclusion
  Plasma balance mean will be calculated with 6 blood samples collected at regular intervals during the visit
The health-related quality (HRQoL) by the self-reported French version of the Short Form (36) Health Survey | Day 1
The health-related quality (HRQoL) by the self-reported French version of the Short Form (36) Health Survey | 3 months after inclusion
The health-related quality (HRQoL) by the self-reported French version of the Short Form (36) Health Survey | 6 months after inclusion
The health-related quality (HRQoL) by the self-reported French version of the Short Form (36) Health Survey | 12 months after inclusion
The health-related quality (HRQoL) by the self-reported French version of the Short Form (36) Health Survey | 18 months after inclusion
The health-related quality (HRQoL) by the self-reported French version of the Short Form (36) Health Survey | 24 months after inclusion
Response to treatment assessed by positron emission tomography-Scan | Day 0
  complete response, partial, stable disease, disease progression
Response to treatment assessed by positron emission tomography-Scan | 6 months after inclusion
  complete response, partial, stable disease, disease progression
Response to treatment assessed by positron emission tomography-Scan | 12 months after inclusion
  complete response, partial, stable disease, disease progression
Response to treatment assessed by positron emission tomography-Scan | 24 months after inclusion
  complete response, partial, stable disease, disease progression
Forgetting to take medication reported by the patient as recorded in a logbook given to the patient | 3 months after inclusion
Forgetting to take medication reported by the patient as recorded in a logbook given to the patient | 6 months after inclusion
Perception of side effect reported by patient as noted in a logbook by the patient | 3 months after inclusion
Perception of side effect reported by patient as noted in a logbook by the patient | 6 months after inclusion
Effect of patients characteristics on plasma balance mean concentration in ibrutinib | 1 months after inclusion
Effect of patients characteristics on plasma balance mean concentration in idelalisib | 1 months after inclusion
Effect of patients genetic polymorphism on plasma balance mean concentration in idelalisib | 1 months after inclusion
Effect of patients therapeutic target DNA polymorphism on treatment response to ibrutinib | Through the completion of study (24 months)
Effect of patients therapeutic target DNA polymorphism on treatment response to idelalisib | Through the completion of study (24 months)
Treatment failure rate in relation with mean concentration of ibrutinib | 1 month after inclusion
Treatment failure rate in relation with mean concentration of idelalisib | 1 month after inclusion
Evaluation of total exposition to ibrutinib (AUCt,ss) with residual concentration at steady state | Through the completion of study (24 months)
Evaluation of total exposition to idelalisib (AUCt,ss) with residual concentration at steady state | Through the completion of study (24 months)
Association of adverse event and quality of life with Short Form (36) Health Survey | Through the completion of study (24 months)
Association of prognostic factors at inclusion and plasma balance mean concentration in ibrutinib | 1 month after inclusion
Association of prognostic factors at inclusion and plasma balance mean concentration in idelalisib | 1 month after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Ysebaert, MD, Principal Investigator — Cancer University Institute of Toulouse Oncopole
Locations (1):
- Cancer University Institute of Toulouse Oncopole, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cadot S, Audebert C, Dion C, Ken S, Dupre L, Largeaud L, Laurent C, Ysebaert L, Crauste F, Quillet-Mary A. New pharmacodynamic parameters linked with ibrutinib responses in chronic lymphocytic leukemia: Prospective study in real-world patients and mathematical modeling. PLoS Med. 2024 Jul 22;21(7):e1004430. doi: 10.1371/journal.pmed.1004430. eCollection 2024 Jul. PMID 39037964
- [Derived] Gallais F, Ysebaert L, Despas F, De Barros S, Dupre L, Quillet-Mary A, Protin C, Thomas F, Oberic L, Allal B, Chatelut E, White-Koning M. Population Pharmacokinetics of Ibrutinib and Its Dihydrodiol Metabolite in Patients with Lymphoid Malignancies. Clin Pharmacokinet. 2020 Sep;59(9):1171-1183. doi: 10.1007/s40262-020-00884-0. PMID 32328976